CLINICAL TRIAL: NCT02542306
Title: Safety and Efficacy of Fibrinogen Concentrate in Aortic Arch Surgery Involving Moderate Hypothermic Circulatory Arrest
Acronym: SEFC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hongjia Zhang (Other)
Collaborators: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor-Investigator, Hongjia Zhang, M.D.Clinical research, Beijing Municipal Science & Technology Commission
Organization: Beijing Municipal Science & Technology Commission (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z141100002114025
Record Dates: First submitted 2015-08-25; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Proximal Aortic Dissection
Keywords: Blood loss; coagulopathy; fibrinogen concentrate; transfusion
MeSH Terms: conditions — Hemorrhage; Hemostatic Disorders | interventions — Fibrinogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fibrinogen concentrate-treated group (Experimental): The initial fibrinogen concentrate dose was 25 - 50 mg/kg, but additional fibrinogen concentrate was administered repeatedly if the first infusion of fibrinogen concentrate did not increase the fibrinogen level over 2.0 g/L.
  Interventions: Drug: fibrinogen concentrate
- non-fibrinogen concentrate-treated group (No Intervention): The participants who did not received fibrinogen concentrate treatment were enrolled as the non-fibrinogen concentrate-treated group

INTERVENTIONS:
Drug: fibrinogen concentrate — Investigators administered fibrinogen concentrate when the plasma fibrinogen level was below 1.5 g/L at 5 minutes after protamine reversal and completion of surgical hemostasis in patients, who comprised the fibrinogen concentrate-treated group.
  Arms: fibrinogen concentrate-treated group

SUMMARY:
Bleeding is a common complication of cardiac surgery, especially aortic arch surgery involving moderate hypothermic circulatory arrest. Fibrinogen concentrate is increasingly used to treat coagulopathic bleeding in cardiac surgery, although its effectiveness and safety are unknown.

Fibrinogen concentrate was administered to 54 patients when the fibrinogen level was below 1.5 g/L after protamine reversal. Additionally, 30 patients were enrolled as the non-FC-treated group.

DETAILED DESCRIPTION:
The aim of this prospective study was to investigate the safety and efficacy of fibrinogen concentrate in patients with acute type A aortic dissection.

Eighty-four acute type A aortic dissection patients undergoing emergency aortic arch surgery involving moderate hypothermic circulatory arrest were included. The clinical data, standard laboratory tests and plasma fibrinogen levels were obtained at 5 time points.

The investigators analyzed the standard laboratory tests, the plasma fibrinogen levels, the volumes of cumulative postoperative drainage and transfused allogenic blood products in 84 patients.

The primary and secondary end points were determined and considered.The primary endpoint (efficacy endpoint) included the volumes of individual allogeneic blood products, volumes of cumulative drainage within 24 h and 48 h and 5 days volumes after infusion of fibrinogen concentrate as well as the rates of reoperation due to bleeding. The secondary endpoint (safety endpoint) for the study was the incidence of serious adverse events from infusion of fibrinogen concentrate to day 45. The serious adverse events defined for the evaluation of safety of fibrinogen concentrate were death, pulmonary embolism and other thromboembolic or ischemic events (myocardial infarction, paraplegia and cerebral infarction).

ELIGIBILITY:
Inclusion Criteria:

* The participants aged 18 years or above who were undergoing emergency aortic arch surgery involving moderate hypothermic circulatory arrest for an acute type A aortic dissection

Exclusion Criteria:

* The participants with congenital or acquired coagulation disorders, previous surgery at the same site, death prior to planned surgery, stroke or myocardial infarction within 2 months before surgery and use of aspirin, clopidogrel or vitamin K antagonists within 2 to 5 days before surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
efficacy endpoint (the volumes of allogeneic blood products, volumes of cumulative drainage within 24 h and 48 h and 5 days | from the time of fibrinogen concentrate administration until the 5th postoperative day
  Investigators hypothesized that the hemostatic therapy with fibrinogen concentrate in acute type A aortic dissection patients resulted in a reduction in the transfusion of allogeneic blood products and drainage volumes compared to the control group that received conventional hemostatic therapy.

SECONDARY OUTCOMES:
safety endpoint (incidence of serious adverse events) | from infusion of fibrinogen concentrate to day 45
  The serious adverse events defined for the evaluation of safety of fibrinogen concentrate were death, pulmonary embolism and other thromboembolic or ischemic events (myocardial infarction, paraplegia and cerebral infarction).

CONTACTS AND LOCATIONS:
Overall Officials: Hongjia Zhang, M.D., Study Chair — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China